CLINICAL TRIAL: NCT00798044
Title: Patient Feedback Effectiveness Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Paul Crits-Christoph, Professor of Psychology in Psychiatry, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: R01DA020799 (NIH); R01DA020799 (NIH); NCT00622154 (obsolete NCT alias)
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Substance Use Disorders
Keywords: quality improvement; feedback; substance use disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Feedback to counselors (Experimental): substance abuse counselors received feedback reports on their average performance and on the average performance of the clinic as a whole. Feedback reports contained information on average alliance, treatment satisfaction, and drug/alcohol use.
  Interventions: Behavioral: Other: quality improvement feedback system; Behavioral: Patient Feedback
- Treatment as Usual (No Intervention): No feedback reports were provided in this arm.

INTERVENTIONS:
Behavioral: Other: quality improvement feedback system — Surveys patients regarding treatment experiences.
  Arms: Feedback to counselors
Behavioral: Patient Feedback — Weekly feedback reports provided to counselors
  Arms: Feedback to counselors

SUMMARY:
The purpose of the study is to determine if a semi-automated quality improvement system that provides addiction counselors with feedback on their average treatment satisfaction and therapeutic alliance (as rated by patients currently in treatment) is superior to no feedback in 32 community-based outpatient addiction treatment clinics.

DETAILED DESCRIPTION:
Quality improvement (Ql) methods are a cornerstone of business and healthcare management throughout the United States yet there have been few studies of Ql interventions in addiction treatment settings. The proposed study tests the effectiveness of one Ql system - Patient Feedback (PF) - at increasing outpatient group therapy attendance and self-reported abstinence. The feasibility and acceptability of PF was established in a six-site study conducted within the National Drug Abuse Treatment Clinical Trials Network. In the proposed study, 32 community-based outpatient treatment programs with approximately 250 clinicians will be randomly assigned to PF, or usual clinic practices. In the PF condition, every week fro 12 weeks clinic patients are invited to complete a 12-item, self-administered survey in which they rate therapeutic alliance and treatment satisfaction, and report past week substance use. These anonymous surveys are faxed by clinic staff to a University of Pennsylvania data center where a custom software application converts the surveys into feedback reports and posts them to a password protected website. Clinicians can access their caseload feedback reports and aggregated reports for the whole clinic; supervisors can only access the aggregated clinic reports. On a monthly basis staff meet as a team to review the feedback reports and develop Ql plans intended to yield improvements in select Ql indicators. The PF website and the monthly PF e-newsletter provide social recognition, clinical resources, and a virtual community for participating clinicians. After 12 weeks, participants in both conditions complete follow-up measures and then both groups are given open access to PF for 12 additional months. During "sustainability phase" staff usage of the PF website is monitored. Alternate versions of the PF Survey are introduced during the sustainability study, including one that monitors HIV risk behavior. The rapid processing of surveys enables near real time feedback to clinic staff. Organizations may share their feedback reports with funding sources, regulatory agencies, policy makers, and other stakeholders. This centralized, semi-automated feedback system eases fulfillment of accreditation requirements and as such, reduces the cost of clinic operations.

ELIGIBILITY:
Inclusion Criteria:

* program: adult, outpatient, non-methadone maintenance substance abuse treatment programs
* clinician: must be leading at least one weekly group with minimum of 5 patients
* must be working at least 20% time at facility

Exclusion Criteria:

* clinics with fewer than 5 clinicians who conduct weekly group counseling
* clinics in which fewer than 50% of clinicians agree to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2006-11; Primary Completion 2008-11 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
clinician average weekly caseload patient-rated therapeutic alliance | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul Crits-Christoph, Ph.D., Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - New York University School of Medicine, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania